CLINICAL TRIAL: NCT02148224
Title: Correlation of Glycemic Index Values and Subjects' Body Composition Parameters
Brief Title: Relationship of Glycemic Index Values and Subjects' Body Composition Parameters
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Nutrifood Research Center, Jakarta, Indonesia (Industry)
Responsible Party: Principal Investigator, Kamalita Pertiwi, Nutrition and Health Science Associate, Nutrifood Research Center, Jakarta, Indonesia
Other Study IDs: 01-NRC-04-2014
Record Dates: First submitted 2014-05-20; First posted 2014-05-28 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Healthy
Keywords: glycemic index; body composition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- healthy without diabetes

SUMMARY:
Glycemic index concept is widely used to determine impact of a food to blood glucose. Although the previous studies showed that glycemic index did not seem to be related with subject-specific factors, currently several studies found conflicting results on the relationship of subjects' characteristics and glycemic index values. This study aims to determine whether body composition parameters, as subject-specific factor, correlate with glycemic index values.

DETAILED DESCRIPTION:
Glycemic index methods are performed according to Food and Agricultural Organization/WHO recommendations.

ELIGIBILITY:
Inclusion Criteria:

* age between 20-40 years
* fasting blood glucose 70-100 mg/dL
* Indonesians

Exclusion Criteria:

* having diabetes
* smoking
* if women, pregnant or lactating
* being allergic to food used in this study
* having gastrointestinal disturbance
* in regular medication
* refusal to sign the consent form

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Study participants will be selected from a group of office workers fulfilling inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2014-04; Primary Completion 2014-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
correlation between glycemic value and body composition | baseline
  Study the correlation between the glycemic values (produced from comparing area under the curve value after ingestion of glucose standard and after consuming test sample) and subjects' body composition parameters: weight, muscle mass, fat mass, percent body fat, BMI, Waist-hip ratio, visceral fat, and estimated trunk fat.
  Pearson's r and its significance value (p-value) will be reported.
glycemic index values of instant noodle | 2 hours postprandial glucose
  The glycemic index is a calculated from measurements of area under the glucose curve after the food is eaten, divided by the corresponding area after the control food is eaten. The value is multiplied by 100 to represent a percentage of the control food.

CONTACTS AND LOCATIONS:
Overall Officials: Kamalita Pertiwi, STP, Principal Investigator — Nutrifood Research Center; Astri Kurniati, MAppSc, Study Chair — Nutrifood Research Center; Lina Antono, MSc, Principal Investigator — Nutrifood Research Center; Susana Susana, MSc, PDEng, Study Chair — Nutrifood Research Center; Mardi Wu, MBA, Study Chair — Nutrifood Research Center
Locations (1):
- Nutrifood Research Center, Propinsi DKI Jakarta, DKI Jakarta, Indonesia

REFERENCES:
- [Background] Carbohydrates in human nutrition. Report of a Joint FAO/WHO Expert Consultation. FAO Food Nutr Pap. 1998;66:1-140. No abstract available. PMID 9743703
- [Background] Srikanthan P, Karlamangla AS. Relative muscle mass is inversely associated with insulin resistance and prediabetes. Findings from the third National Health and Nutrition Examination Survey. J Clin Endocrinol Metab. 2011 Sep;96(9):2898-903. doi: 10.1210/jc.2011-0435. Epub 2011 Jul 21. PMID 21778224
- [Background] Mettler S, Lamprecht-Rusca F, Stoffel-Kurt N, Wenk C, Colombani PC. The influence of the subjects' training state on the glycemic index. Eur J Clin Nutr. 2007 Jan;61(1):19-24. doi: 10.1038/sj.ejcn.1602480. Epub 2006 Jul 12. PMID 16835599